CLINICAL TRIAL: NCT01063348
Title: A Double-Blind, Placebo-Controlled Study of N-Acetyl Cysteine in Pathologic Skin Picking
Brief Title: N-Acetyl Cysteine in Pathologic Skin Picking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010PSPNAC
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Pathologic Skin Picking; Neurotic Excoriation; Psychogenic Excoriation; Dermatillomania
Keywords: N-Acetyl Cysteine; Picking; Impulse Control Disorder; Obsessive Compulsive Disorder
MeSH Terms: conditions — Excoriation Disorder; Disruptive, Impulse Control, and Conduct Disorders; Obsessive-Compulsive Disorder | interventions — Acetylcysteine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetyl Cysteine (Active Comparator): N-Acetyl Cysteine - 600mg tablets by mouth (dosing 1200mg - 3000mg qd)
  Interventions: Drug: N-Acetyl Cysteine
- Placebo (Placebo Comparator): Matching placebo taken daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetyl Cysteine — Week 0 (Visit 1) - Week 3 (V2): 1200mg/day (600mg po qam and 600mg po qpm) Week 3 (V2) - Week 6 (V3): 2400mg/day (1200mg po qam and 1200mg po qpm) Week 6 (V4) - Week 12 (V5): 3000mg/day (1200mg po qam and 1800mg po qpm)
  Other Names: NAC
  Arms: N-Acetyl Cysteine
Drug: Placebo — Matching placebo capsules taken in same amount of pills as the active medication.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The goal of the proposed study is to evaluate the comparative efficacy of N-acetyl cysteine to placebo in pathologic skin picking. Thirty subjects with pathologic skin picking will receive 12 weeks of double-blind treatment with N-acetyl cysteine or matching placebo. The hypothesis to be tested is that N-acetyl cysteine will be more effective than placebo in patients with pathologic skin picking. The proposed study will provide needed data on the treatment of an often disabling disorder that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
Pathologic skin picking involves repetitive, ritualistic, or impulsive picking of otherwise normal skin leading to tissue damage, personal distress, and impaired functioning. Although skin picking has been described in the medical literature for over one-hundred years, it remains a poorly understood psychiatric issue and often goes undiagnosed and untreated.

Picking behavior does not by itself suggest a psychiatric disorder. Pathology exists in the focus, duration and extent of the behavior, as well as the reasons for picking, associated emotions, and resulting problems. Patients with PSP report thoughts of picking or impulses to pick that are irresistible, intrusive and/or senseless. These thoughts, impulses, or behaviors also cause marked distress for patients and significantly interfere with other activities. Unlike normal picking behavior, the pathologic form of skin picking is recurrent and usually results in noticeable skin damage.

Thirty subjects with pathologic skin picking will receive 12 weeks of double-blind treatment with N-acetyl cysteine or matching placebo. The hypothesis to be tested is that N-acetyl cysteine will be more effective than placebo in patients with pathologic skin picking. The proposed study will provide needed data on the treatment of an often disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-65;
2. Current diagnosis of pathologic skin picking as determined by criteria proposed by Arnold et al. (2001) for at least 6 months duration

Exclusion Criteria:

1. Unstable medical illness or clinically significant abnormalities on prestudy laboratory tests or physical examination;
2. History of seizures;
3. Myocardial infarction within 6 months;
4. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
5. Need for medication other than NAC with possible psychotropic effects or unfavorable interactions with NAC;
6. Clinically significant suicidality (score or 3 or 4 on item 3 of the Hamilton Depression Rating Scale);
7. Lifetime history of DSM-IV bipolar disorder type I, dementia, or schizophrenia or any other DSM-IV psychotic disorder;
8. Current or recent (past 3 months) DSM-IV substance abuse or dependence;
9. Illegal substance use within 2 weeks of study initiation;
10. Initiation of pharmacotherapy, psychotherapy, or behavior therapy from a mental health professional within 3 months prior to study baseline for the treatment of pathologic skin picking;
11. Previous treatment with N-acetyl cysteine;
12. Treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline;
13. Asthma (given possible worsening of asthma due to NAC)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Arnold LM, Auchenbach MB, McElroy SL. Psychogenic excoriation. Clinical features, proposed diagnostic criteria, epidemiology and approaches to treatment. CNS Drugs. 2001;15(5):351-9. doi: 10.2165/00023210-200115050-00002. PMID 11475941
- [Background] Grant JE, Odlaug BL. Update on pathological skin picking. Curr Psychiatry Rep. 2009 Aug;11(4):283-8. doi: 10.1007/s11920-009-0041-x. PMID 19635236
- [Derived] Grant JE, Chesivoir E, Valle S, Ehsan D, Chamberlain SR. Double-Blind Placebo-Controlled Study of Memantine in Trichotillomania and Skin-Picking Disorder. Am J Psychiatry. 2023 May 1;180(5):348-356. doi: 10.1176/appi.ajp.20220737. Epub 2023 Feb 22. PMID 36856701
- [Derived] Grant JE, Chamberlain SR, Redden SA, Leppink EW, Odlaug BL, Kim SW. N-Acetylcysteine in the Treatment of Excoriation Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 May 1;73(5):490-6. doi: 10.1001/jamapsychiatry.2016.0060. PMID 27007062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-Acetyl Cysteine | Placebo
Started | 35 | 31
Completed | 32 | 21
Not Completed | 3 | 10
Not completed — Lost to Follow-up | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetyl Cysteine | Placebo | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (11.6) | 34.7 (10.5) | 34.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 58
  Male | 2 | 6 | 8
Any Psychiatric Comorbidity [Number; unit: participants]
  Yes | 20 | 14 | 34
  No | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale (YBOCS) Modified for PSP (NE-YBOCS)
Description: The entire study for an individual subject will last 12 weeks. Every 3 weeks the subject will take the YBOCS for the duration of the 12 weeks. At each of these visits the outcome will be assessed.
  The minimum score is 0 and the maximum score is 40, with a higher score being more severe skin picking. There are two sub-scales: one for urges (ranges from 0 to 20) and one for behaviors (ranges from 0 to 20). The total of the scores of each of the sub-scales is the total YBOCS score. That is what will be reported.
Time Frame: Once every three weeks during the 12 week study for each subject
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetyl Cysteine | Placebo
Number analyzed (Participants) | 32 | 21
units on a scale
  Baseline | 18.8 (5.3) | 17.6 (4.8)
  Week 3 | 16.1 (5.9) | 17.3 (5.4)
  Week 6 | 13.9 (6.3) | 16.3 (6.9)
  Week 9 | 12.4 (5.8) | 15.0 (7.4)
  Week 12 | 11.5 (5.4) | 14.1 (7.5)

2. Secondary Outcome: Skin Picking Self Assessment Scale (SP-SAS)
Description: The entire study for an individual subject will last 12 weeks. Every 3 weeks the subject will take the YBOCS for the duration of the 12 weeks. At each of these visits the outcome will be assessed.
  The minimum score is 0 and the maximum score is 48 with higher scores meaning more severe skin picking. The total of all of the questions equals the total reported SP-SAS score.
Time Frame: Once every three weeks for the duration of the 12 week study for each subject
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetyl Cysteine | Placebo
Number analyzed (Participants) | 32 | 21
units on a scale
  Baseline | 28.6 (6.2) | 28.6 (7.0)
  Week 3 | 24.8 (7.2) | 25.5 (6.2)
  Week 6 | 21.9 (8.0) | 25.0 (8.8)
  Week 9 | 21.5 (10.3) | 24.2 (8.5)
  Week 12 | 19.4 (8.7) | 24.5 (9.0)

ADVERSE EVENTS:
Arm/Group | N-Acetyl Cysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 9/35 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-Acetyl Cysteine (N=35) | Placebo (N=31)
Nausea (Gastrointestinal disorders) | 5 | 1
Dry Mouth (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dizziness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No